CLINICAL TRIAL: NCT02237131
Title: Continuous Versus Cyclic Use of Oral Contraceptives Following Surgery for Symptomatic Endometriosis
Brief Title: Continuous Versus Cyclic Oral Contraceptives for Endometriosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Nikos Vlahos, M.D, F.A.C.O.G Ass. Professor of Gynecology and Obstetrics, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: NV04042013
Record Dates: First submitted 2014-03-22; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Dysmenorrhea; Pelvic Pain; Dyspareunia; Endometrioma
Keywords: Endometriosis; Oral contraceptives; Laparoscopy
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain; Dyspareunia; Endometriosis | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral contraceptives cyclic (Experimental): Oral contraceptives containing 0.03 mg ethinyl estradiol and 3mg drospirenone will be administered. One tablet a day for 21 days followed by 7 days pill free. The regimen will be repeated for the duration of the trial.
  Interventions: Drug: Oral contraceptives cyclic; Drug: Oral contraceptives continuous
- Oral contraceptives continuous (Active Comparator): Oral contraceptives containing 0.030 mg ethinyl estradiol and 3mg drospirenone will be administered. One tablet a day for the duration of the trial.
  Interventions: Drug: Oral contraceptives cyclic; Drug: Oral contraceptives continuous

INTERVENTIONS:
Drug: Oral contraceptives cyclic — tables containing Ethinyl estradiol 0.03mg and drospirenone 3mg will be administered in a cyclic fashion 21 days on 7 days off pill for 6 cycles.
  Other Names: Yasmin.
Drug: Oral contraceptives continuous — Patients will be treated with oral contraceptives containing 0.03mg ethinyl estradiol and 3 mg drospirenone per day in a continuous fashion.
  Other Names: Yasmin

SUMMARY:
To evaluate the efficacy of oral contraceptives in a continuous fashion versus the usual cyclic fashion in the recurrence of endometriosis related symptoms and endometriomas following fertility-sparing surgery.

DETAILED DESCRIPTION:
Oral contraceptives containing 0.03 mg ethinyl estradiol and 3mg drospirenone will be administered. One tablet a day for 21 days followed by 7 days pill free (cyclic fashion) or one tablet a day in a continuous fashion.

ELIGIBILITY:
Inclusion Criteria:

Women of reproductive age with Symptomatic endometriosis following fertility sparing surgery

Exclusion Criteria:

Contraindications of use of oral contraceptives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain | 6 months
  In each visit patients will complete a detailed 25-item self-administered questionnaire (www.endometriosisfoundation.org/WERF-WHSS-Questionnaire-English.pdf) related to the presence of pelvic pain (scoring of pelvic pain)

SECONDARY OUTCOMES:
recurrence rate for endometrioma | 6 months
  Physical and transvaginal sonographic examination

OTHER OUTCOMES:
dysmenorrhea | 6 months
  In each visit patients were asked to complete a detailed 25-item self-administered questionnaire (www.endometriosisfoundation.org/WERF-WHSS-Questionnaire-English.pdf) related to the presence of dysmenorrhea (scoring of dysmenorrhea)

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Vlahos, AssProfessor, Study Chair — University of Athens, 2nd Department of Obstetrics and Gynecology; Olga Triantafyllidou, MD, Principal Investigator — University of Athens, 2nd Department of Obstetrics and Gynecology
Locations (1):
- Aretaieion Hospital, Athens, Athens, Greece